CLINICAL TRIAL: NCT06051331
Title: The Effect of Simulation-Based Breast Health Education on Breast Cancer Awareness and Breast Self-Examination Practices of Afgan Refugee Women: A Randomized Control Trial
Brief Title: The Effect of Simulation-Based Breast Health Education on Breast Cancer Awareness and Breast Self-Examination Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nilgun Kuru Alici, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D69071
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Health Knowledge, Attitudes, Practice
Keywords: Afghan; Breast Cancer; Awareness; Health Education
MeSH Terms: conditions — Breast Neoplasms; Behavior; Health Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Simulation-based breast health education
  Interventions: Behavioral: simulation-based breast health education
- Control group (No Intervention): The control group will not take part the simulation-based breast health education

INTERVENTIONS:
Behavioral: simulation-based breast health education — The intervention group will receive simulation-based breast health education once a week for eight weeks. The simulation- based breast health education program will compose two part. The first part, it will theoretical education and second part will continue as practical education. On the plan date, a 60-min lecture will give about breast cancer, its risk factors, interventions to reduce the risk of breast cancer, the value of early diagnosis and cancer screening. After a 10-min break, course attendees watched a 20-min video, after which the course attendees' questions will answer.
  Arms: Experimental group

SUMMARY:
This study aimed to evaluate the effect of simulation-based breast health education on breast cancer awareness and breast self-examination practices of Afghan refugee women. The study hypothesized that simulation-based breast health education would have an effect on breast cancer awareness and breast self-examination practices scores among Afghan refugee women.

DETAILED DESCRIPTION:
Purpose: The aim of the research is to examine the effects of simulation-based breast health education on breast cancer awareness and breast self-examination practices of Afghan refugee women.

Methods: The study will conduct with 64 (32 in the intervention group, and 32 in the control group) Afghan. The study population consisted of Afghan women. The simulation-based breast health education will applied to the intervention group once a week for 8 weeks.

No intervention will offer to the control group. Data will collected by a socio-demographic questionnaire, Breast Cancer Awareness Measure (BCAM) and breast self-examination practices checklist.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years,
* must be able to speak Turkish or Dari.

Exclusion Criteria:

* breast cancer

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
The Breast Cancer Awareness Measure Score | up to 8 weeks
  The Breast Cancer Awareness Measure was developed by the Cancer Research UK group of Kings College London in 2009.It is a questionnaire that assesses seven domains of Breast Cancer (BC) awareness: knowledge of BC symptoms, breast self-examination, confidence of noticing a change in the breasts, age and lifetime risk of Breast Cancer, urgency if a change in breast is noticed, BC risk factors, and Breast Cancer screening. In this study, Dari version of The Breast Cancer Awareness Measure which was translated from English into Dari by an official translator. The respondent receives 1 point if they can correctly identify at least 5 signs of breast cancer, 1 point if they select the oldest woman for the age-related risk item, and 1 point if they report performing breast examination once a month. Incorrect answers receive 0 points. The total score is between 0 and 3 and there is no cut-off point.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Kuru Alici N, Arikan Donmez A, Aktas O, Zeytun Z. The effect of simulation-based breast health education on breast cancer awareness and breast self-examination skills of Afghan refugee women: a randomized controlled trial. BMC Public Health. 2025 Jun 2;25(1):2048. doi: 10.1186/s12889-025-23313-y. PMID 40457306